CLINICAL TRIAL: NCT04569006
Title: Level of Agreement in the Assessment of Carotid Plaque Composition Between Multi-contrast and Multi-sequence MRI
Brief Title: Multi-contrast Versus Multi-sequence Carotid MRI
Status: Recruiting | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: ABR73156
Record Dates: First submitted 2020-09-16; First posted 2020-09-29 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Atherosclerosis
MeSH Terms: conditions — Atherosclerosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Carotid plaque tissue retrieved only from patients undergoing carotid endarterectomy for regular patient care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The objective of this study is to validate 2 multi-contrast sequences, namely the Multi-contrast ATherosclerosis Characterization (MATCH) and Bright-blood and black-blOOd phase SensiTive (BOOST) inversion recovery sequence for the quantification of atherosclerotic plaque components with conventional multi-sequence MRI and histology.

DETAILED DESCRIPTION:
Rationale: Rupture of a vulnerable atherosclerotic plaque is the most important cause of stroke and myocardial infarction. Magnetic Resonance Imaging (MRI) with its high soft tissue contrast is well suited for atherosclerotic plaque imaging to identify high-risk plaques. High soft tissue contrast enables the visualisation of different plaque components based on which the plaque can be classified as stable or vulnerable. To identify the various plaque components, in a conventional MRI examination multiple MRI sequences are acquired, which can take approximately 30-40 minutes. This can be uncomfortable for the patient and it is impractical in daily clinical practice. As an alternative, multi-contrast sequences have recently been developed which acquire multiple contrast weightings simultaneously, significantly reducing the scan time (< 6 minutes). Apart from a reduction in scan time, because these contrast weightings are acquired simultaneously, they are inherently co-registered which is not the case with conventional sequences.

Objective: The objective of this study is to validate 2 multi-contrast sequences, namely the Multi-contrast ATherosclerosis Characterization (MATCH) and Bright-blood and black-blOOd phase SensiTive (BOOST) inversion recovery sequence for the quantification of atherosclerotic plaque components with conventional multi-sequence MRI and histology.

Study design: cross-sectional validation study Study population: 40 patients with a carotid artery plaque ≥2 mm based on ultrasound or Computed Tomography Angiography.

Intervention (if applicable): not applicable Main study parameters/endpoints: the presence and volumetric measures of plaque components (fibrous tissue, lipid-rich necrotic core, intraplaque hemorrhage and calcifications) and volumetric measures of the vessel wall and lumen as assessed with multi-contrast MRI will be compared to those as assessed by conventional multisequence MRI and, if available, histology of the surgically removed specimen in patients that are scheduled for carotid endarterectomy.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, a subject must meet the following criteria:

* Patients with a carotid plaque ≥ 2 mm thick based on ultrasound or CTA
* Age 18 years or older (no maximum age)
* Informed consent by signing informed consent form regarding this study

Exclusion Criteria:

A potential subject who meets any of the following criteria will be excluded from participation in this study:

* Patients with carotid plaque ≤ 2 mm in size based on ultrasound or CTA
* Standard contra-indications for MRI (electronic implants like pacemakers or other electronic implants, metallic eye fragments, vascular clips, claustrophobia, etc.)
* Severe co-morbidity, dementia or pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 40 patients (18 years or older) with a carotid plaque ≥ 2 mm based on ultrasound or CTA, will be included in this study. These patients will undergo a 3T MRI scan. Inclusion will be done by an investigator. All the research will take place at Maastricht University Medical Centre (MUMC). Vascular surgeons, neurophysiologists and neurologists at MUMC are willing to participate in this study. Some of the included patients will be scheduled for CEA as part of standard clinical care. The MRI scan of these patients will take place at least one day before CEA is performed. At MUMC, approximately 10 patients per month fit the criteria (≥ 2 mm carotid plaque size).
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2021-04-08 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Presence of Intra Plaque Hemorrhage (IPH) | through study completion, an average of 6 months
  The primary objective is to investigate the level of agreement between scoring presence of IPH on MR images acquired with MP-RAGE (conventional sequence) with scoring IPH on the multi-contrast sequences. The level of agreement will be assessed by calculating Cohen's k.

SECONDARY OUTCOMES:
Scoring the presence of other plaque tissues | through study completion, an average of 6 months
  In addition, we will report the sensitivity and specificity of scoring the presence of IPH, a LRNC, calcifications, a thin or rupture fibrous cap, and ulcerations using the multi-contrast images with the scores based on the conventional multi-sequence images as reference standard.
Calculate correlation between plaque tissues | through study completion, an average of 6 months
  To study the correlation between the vessel wall and luminal volume and volumes of calcifications, LRNC and IPH as delineated on the multi-contrast sequences versus the conventional multisequence MRI protocol.
Correlation between plaque tissues components and histology | through study completion, an average of 6 months
  To study the correlation between the presence/volume of calcifications, LRNC, thin or ruptured fibrous cap, ulcerations and IPH as quantified using the multi-contrast MRI sequences and histology.

CONTACTS AND LOCATIONS:
Locations (1):
- Maastricht University Medical Center, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No